CLINICAL TRIAL: NCT02216604
Title: Physical Activity Intervention Program for Childhood Cancer Patients Under Chemo- and/or Radiation Therapy
Brief Title: Exercise in Pediatric Cancer Patient Undergoing Anti-Cancer Treatment
Acronym: ONKOKIDS-HD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Cancer Research Center (Other)
Collaborators: University Hospital Heidelberg (Other); Heidelberg University (Other); University of Leipzig (Other); Children's Medical Hospital, University of Leipzig, Leipzig, Germany (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: S105-2011
Record Dates: First submitted 2014-08-13; First posted 2014-08-15 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Childhood Cancer
Keywords: Exercise; Pediatric oncology; Physical Performance; Quality of Life; Feasibility; during primary; anticancer treatment
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Multimodal Exercise intervention (console-based training, age-specific resistance training and body awareness)
  Interventions: Behavioral: Multimodal Exercise Intervention
- Control (No Intervention): age, disease and gender matched

INTERVENTIONS:
Behavioral: Multimodal Exercise Intervention — During their inpatient hospitalization the participants perform 3-5x weekly guided training sessions about 15-30min. The intervention includes: game console-based training using Nintendo Wii® (endurance, strength endurance and balance), age-specific resistance training and sessions of body awareness. During the outpatient phases the participants perform a home-based exercise training 3-5x weekly using a training manual. In addition, the patients obtain a movement diary and a pedometer for documenting their activity level.
  Arms: Intervention group

SUMMARY:
Today about 80% childhood cancer patients become long-time survivors. In spite of the high cure rates the diagnosis cancer is associated with a variety of disease and treatment-related psychological and physical impairments mostly present into adulthood. So the attention has to focus on the improvement of these problems such as motor limitation, dysfunction of the cardiovascular system, reduced muscle strength, overweight, osteoporosis and diminished quality of life (Qol). Although exercisel intervention studies in this field are generally scarce, the results of these studies are promising. Up to now studies during the acute phase of treatment are missing almost completely. The aim of this feasibility study is to evaluate the potential benefits of a modular exercise intervention program for childhood cancer patients startunf in parallel with treatment and longlasting for one year. Across two years cancer patients of the Children's Hospital of the University Clinic of Heidelberg aged 5-21 years, free of any contraindications for physical activity will be recruited. All participants are asked to complete a physical assessment battery (strength, endurance and balance capacity, posture control, functional mobility, range of motion) and additionally two questionnaires concerning Qol and motivation, at baseline and every three months following one year

ELIGIBILITY:
Inclusion Criteria:

* pediatric cancer diagnosis (primary leukemia, brain tumors and bone tumors
* date of diagnosis not longer than 8 weeks ago

Exclusion Criteria:

* severe cardiac impairment
* bone metastasis inducing skeletal fragility
* other orthopedic diseases or any other circumstance that would impede ability to give informed consent or adherence to study requirements.

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2011-05; Primary Completion 2018-12 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Feasibility after 6 month | after primary treatment (6 month)
  Will be measured as the proportion of patients following the exercise prescription.

SECONDARY OUTCOMES:
Physical performance | after primary treatment (6 month) and after one year
  Strength (handheld dynamometer), endurance and balance capacity (TUDS, one leg stand), postural control functional mobility (posturomed & force plate), range of motion (goniometer)
Quality of Life | after primary treatment (6 month) and after one year
  KINDL questionnaire
Feasibility between 6 and 12 month | between end of primary treatment (6 month) and one year
  Will be measured as the proportion of patients following the exercise prescription.

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Wiskemann, PhD, Principal Investigator — National Center for Tumor Diseases
Locations (1):
- Children's Hospital of the University Hospital of Heidelberg, Heidelberg, Germany